CLINICAL TRIAL: NCT02453698
Title: Stimulant Effects on Brain Activity During the Stop Signal Task
Brief Title: Stimulant Effects on Brain Activity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Russell Schachar, Staff Physician, The Hospital for Sick Children
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1000020845
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Last update posted 2015-05-25 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Volunteers
Keywords: Stop task; modulatory effect of MPH; bottom-up and top-down; cognitive processes
MeSH Terms: interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Methylphenidate (Experimental)
  Interventions: Drug: Methylphenidate
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate — oral dose of methylphenidate. The MPH dose was selected based on previous studies in healthy adults (Mehta et al., 2000; Volkow, Fowler, Wang, Ding, & Gatley, 2002) and adults with ADHD (Aron et al., 2003). MPH reaches its peak plasma concentration 1-3 hours after an oral dose, and has a plasma half-life of 1.5-2.5 hours.
  Arms: Methylphenidate
Other: Placebo — Lactose Placebo
  Arms: Control Group

SUMMARY:
The aim of this study is to investigate the effects of Methylphenidate on neural activity underlying inhibitory control and error monitoring in healthy adults. More specifically, the investigators aim to establish the baseline modulatory effect of Mehtlylphenidate on bottom-up and top-down aspects of these cognitive processes. This work will further our understanding of Attention Deficit Hyperactivity Disorder, Methylphenidate, and executive functioning.

DETAILED DESCRIPTION:
Methylphenidate (MPH) is the stimulant medication most commonly used in the treatment of attention deficit hyperactivity disorder (ADHD). MPH suppresses the reuptake of dopamine by blocking dopamine transporter, which is elevated in ADHD. However, the precise mechanism by which suppressed dopamine transporter activity relieves ADHD symptoms is not fully understood, partly because dopamine pathways are implicated in various processes that could play a role in the deficits of ADHD and other disorders. MPH-induced dopamine variation has extensive effects in the brain and influences various executive functions in unknown ways.

Hypotheses:

Inhibitory Control: The investigators predict that MPH should increase the top-down activity in right dorsolateral prefrontal cortex associated with response restraint during go-phases and bottom-up activity in caudate and right inferior frontal cortex associated with response cancellation during successful stop trials. A greater modulation of top-down or bottom-up activity would imply a selective effect of MPH on one pathway over the other.

Error Processing: The investigators predict that MPH should increase the intensity of deactivation in the bottom-up dopamine pathway on error detection (substantia nigra, dorsal striatum and ACC), and increase the intensity of deactivation in the top-down pathway on post-error slowing (caudal OFC, ventral striatum, ventral substantia nigra). A greater modulation of top-down or bottom-up activity would imply a selective effect of MPH on one pathway over the other.

ELIGIBILITY:
Inclusion Criteria

* Healthy, non-smoking, male and female volunteers, between 18 to 35 years of age inclusive, right-handed
* Body Mass Index that is within 18.5-29.9 kg/m2, inclusive
* Healthy, according to the medical history, vital signs, and physical examination (within 2 years prior to study enrollment)
* Systolic blood pressure between 100-140 mmHg, inclusive, and diastolic blood pressure between 60-90 mmHg, inclusive, and heart rate between 50-100 bpm, inclusive, unless deemed not clinically significant by the Principal Investigator/ Sub-Investigator?
* Capable of giving written informed consent prior to receiving any study medication
* Female subjects must fulfill at least one of the following:

  * Agree to avoid pregnancy and use medically acceptable method of contraception from at least 30 days prior to the study, during the study, and until 30 days after the study has ended (last study procedure). Medically acceptable methods of contraception include oral contraceptives, hormonal patch, implant or injection intrauterine device, or double barrier method (condom with foam or vaginal spermicidal suppository, diaphragm with spermicide). Complete abstinence alone can be used as a method of contraception.
  * Be surgically sterile for a minimum of 6 months
  * Post-menopausal for a minimum of 1 year

Exclusion Criteria

* Known history or presence of any clinically significant hepatic (e.g. hepatic necrosis, jaundice, hepatobiliary disease), renal, gastrointestinal (e.g. peptic ulcer), cardiovascular (e.g. angina, myocardial infarction), cerebrovascular, pulmonary, endocrine (e.g. diabetes, hypophosphatemia), immunological, musculoskeletal (e.g. rhabdomyolysis, myopathy), neurological, psychiatric, dermatological, or hematological disease or condition
* Presence of any clinically significant illness within 30 days prior to dosing
* Presence of any significant physical or organ abnormality
* Known history or presence of:

  * Alcohol abuse or dependence within one year prior to drug administration
  * Drug abuse or dependence
  * Hypersensitivity to methylphenidate or other medications
  * Gout
  * Food allergies and/or presence of any dietary restrictions
  * Severe allergic reactions (e.g. anaphylactic reactions, angioedema)
* Participation in another clinical trial or receiving an investigational drug within 30 days of the study commencement or during the study
* Use of any prescription medication within 14 days prior to drug administration (except for hormonal contraceptives)
* Use of any over-the-counter medications (including herbal and/or dietary supplements and/or teas) within 14 days prior to drug administration (except for spermicidal/barrier contraceptive products)
* Any major surgery within 6 months prior to the start of the study
* Pregnant or lactating
* Lactose intolerance
* Contraindication for MRI (using hospital's standard screening procedure)
* Smoking

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Neural activity assessed using fMRI | 7 days
  Assessed using fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Russell Schachar, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada